CLINICAL TRIAL: NCT00382928
Title: Automatic External Defibrillation Monitoring in Cardiac Arrest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Foundation for Atlanta Veterans Education and Research, Inc. (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, A. Maziar Zafari, Chief, Cardiology, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1216-2004
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular
Keywords: Randomized Controlled Trials; Defibrillators; Medical Devices
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Group (No Intervention): Patients will receive standard of care measures in case of cardiac arrest. They will not receive AECD monitoring or intervention
- AECD Monitoring + Standard of Care Group (Experimental): Patients will receive AECD monitoring and intervention in addition to standard of care in case of cardiac arrest during admission to the hospital. Defibrillation of pulseless VT/VF by AECD.
  Interventions: Device: Defibrillation of pulseless VT/VF by AECD

INTERVENTIONS:
Device: Defibrillation of pulseless VT/VF by AECD — In case of cardiac arrest caused by shockable rhythms the automatic external cardioverter defibrillator (AECD) will automatically deliver defibrillation. Automated External Cardioverter Defibrillator (AECD; The PowerHeart CRM, Cardiac Science Inc., Seattle, WA) is a device attached to the chest wall by pads, monitors the electrocardiogram, and is capable of automatically delivering electric countershock to appropriate rhythms without operator intervention. The device will deliver only one shock of 150 Joules for pulseless ventricular tachycardia and ventricular fibrillation.
  Arms: AECD Monitoring + Standard of Care Group

SUMMARY:
We propose to randomize automatic external cardioverter/defibrillators (AECD) in patients who are at high risk for life-threatening abnormal heart rhythms (arrhythmias) and are admitted to the telemetry ward, all other treatments being constant including cardiopulmonary resuscitation.

We hypothesize that the automatic, rapid, accurate and specific diagnostic and therapeutic technology used in AECDs will further increase the rate of survival in patients with cardiac arrest through rapid and automatic defibrillation, independent of operator initiation, as compared to standard cardiopulmonary resuscitation initiated by healthcare providers.

DETAILED DESCRIPTION:
Cardiac arrest (CA) is defined as the sudden cessation of effective cardiac pumping function as a result of either ventricular asystole (inactivity of the heart) or pulseless ventricular tachycardia/ventricular fibrillation (VT/VF). Pulseless ventricular tachycardia/ventricular fibrillation is an abnormal electrical activity of the ventricles of the heart. Rapid diagnosis and treatment are essential because first, more than a few minutes of total CA results in permanent damage to the brain due to lack of oxygen, and second, the success of resuscitative measures is related to the rapidity with which they are instituted following arrest. For a person in VT/VF the probability of successful defibrillation and subsequent survival to hospital discharge is directly and negatively related to the interval between onset of VT/VF and delivery of first shock.

Comparison: By using AECDs we will evaluate if an automatic, rapid, accurate and specific diagnostic technology will further increase the rate of survival in patients with VT/VF by rapid and automatic defibrillation, independent of operator initiation, as compared to standard cardiopulmonary resuscitation (CPR) with conventional defibrillators initiated by healthcare providers. This trial will be a randomized, controlled trial and will test if AECDs can improve outcome measures when compared to traditional responses.

Conventional defibrillators are manually operated defibrillators that have to be attached to the patient and operated by a healthcare provider or layperson. In contrast, the purpose of AECDs is to automatically detect life-threatening arrhythmias and deliver external shocks according to a programmable prescription for hospitalized patients, who may be at transient risk for the development of life-threatening arrhythmias. AECDs immediately and automatically monitor, detect and treat cardiac arrhythmias with no human intervention. The AECD proposed to be utilized in this trial, PowerHeart CRM, a product of Cardiac Science, Inc, has been evaluated in the hospital setting to assess safety and efficacy, and has been approved by the FDA to be prophylactically attached to hospital patients and provide automatic defibrillation therapy without human intervention.

All patients admitted to the telemetry unit will be asked to volunteer for this study. Up to 3,000 patients will be asked to volunteer in this study during their stay in the telemetry unit. This study will evaluate if there is a way to improve survival in CA by comparing two groups

Group 1: This group includes patients admitted to telemetry unit who will undergo standard measures of CPR in case cardiac arrest is suspected.

Group 2: This group includes patients admitted to telemetry unit who will have an AECD attached to the chest wall and who will also undergo standard measures of CPR in case of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to telemetry ward and emergency department
* Age > 18 years.

Exclusion Criteria:

* Pregnant women
* Patients with R wave less than 0.5 millivolts.
* Patients with functioning Internal Cardiac Device.
* Patients with cardiac pacemakers if oversensing by AECD is demonstrated (double counting of pacer spikes).
* Patients with visible chest lesions that would prevent AECD pad placement.
* Patients who are designated Do Not Resuscitate.
* Right bundle branch block.
* Patients with Parkinson's disease.
* Patients with seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Maziar Zafari, M.D., Ph.D, Principal Investigator — Division of Cardiology, Atlanta Veterans Adminstration Medical Center/ Emory University, Decatur, GA
Locations (1):
- Atlanta Veterans Adminstration Medical Center, Decatur, Georgia, United States

REFERENCES:
- [Derived] Ali B, Bloom H, Veledar E, House D, Norvel R, Dudley SC, Zafari AM. Automated external cardioversion defibrillation monitoring in cardiac arrest: a randomized trial. Trials. 2008 Jun 11;9:36. doi: 10.1186/1745-6215-9-36. PMID 18547438
- See also: Click here for detailed information about this study: Automated external cardioversion defibrillation monitoring in cardiac arrest: a randomized trial — http://www.trialsjournal.com/content/9/1/36

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and ninety two patients were recruited in the time period between 10/10/2006 to 7/20/2007 to the telemetry ward of the Atlanta VA Medical Center.
Groups:
- No Intervention: Standard of Care Group: Patients will receive standard of care measures in case of cardiac arrest. They will not receive AECD monitoring or intervention
- Experimental: AECD Monitoring + Standard of Care Group: Patients will receive AECD monitoring and intervention in addition to standard of care in case of cardiac arrest during admission to the hospital.
Period: Overall Study
Arm/Group | No Intervention: Standard of Care Group | Experimental: AECD Monitoring + Standard of Care Group
Started | 97 | 95
Completed | 97 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention: Standard of Care Group | Experimental: AECD Monitoring + Standard of Care Group | Total
Number analyzed (Participants) | 97 | 95 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 95 | 192
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (3.4) | 61.7 (3.4) | 61.9 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 94 | 92 | 186
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 2 | 2
  White | 53 | 42 | 95
  Black | 44 | 51 | 95
Clinical Characteristics of Study Subjects [Number; unit: participants]
  History of Heart Failure | 20 | 25 | 45
  New Diagnosis of Heart Failure | 4 | 6 | 10
  Diabetes mellitus | 35 | 46 | 81
  History of Coronary Artery Disease | 42 | 35 | 77
  Hypertension | 74 | 79 | 153
  Hyperlipidemia | 53 | 55 | 108
EKG on admission [Number; unit: participants]
  normal sinus rhythm | 81 | 84 | 165
  Atrial fibrillation/flutter | 11 | 9 | 20
  supraventricular tachycardia | 2 | 0 | 2
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Defibrillation
Description: Time to defibrillation: interval between onset of VT/VF and delivery of first shock. Expected time to defibrillation for AECD group: 30±30 seconds; expected time to defibrillation for Standard of Care group: 180±180.
Time Frame: 10 minutes
Population: There was only one patient in the Intervention group who received defibrillation.
  No patients had CPR or defibrillation in the standard of care group.
Measure: Number; unit: participants
Groups:
- Experimental: AECD Monitoring + Stand of Care Group: Patients will receive AECD monitoring and intervention in addition to standard of care in case of cardiac arrest during admission to the hospital.
Arm/Group | Experimental: AECD Monitoring + Stand of Care Group | No Intervention: Standard of Care Group
Number analyzed (Participants) | 95 | 97
participants | 94 (50) | 97

2. Secondary Outcome: Frequency of Abnormal Rhythms Monitored by the AECD
Time Frame: During the duration of hospital admission on the telemetry ward.
Population: Only the AECD+Standard of Care Group was monitored in this portion of the study.
Measure: Number; unit: participants
Groups:
- AECD Monitoring + Standard of Care Group: Patients will receive AECD monitoring and intervention in addition to standard of care in case of cardiac arrest during admission to the hospital.
- Standard of Care: Patients will receive standard of care measures in case of cardiac arrest. They will not receive AECD monitoring or intervention.
Arm/Group | AECD Monitoring + Standard of Care Group | Standard of Care
Number analyzed (Participants) | 95 | 0
participants
  Atrial Fibrillation/Flutter | 9 |
  Supraventricular Tachycardia | 1 |
  Premature Ventricular Complexes | 10 |
  Non-Sustained Ventricular Tachycardia | 5 |

3. Secondary Outcome: Survival to Discharge
Time Frame: At discharge
Measure: Number; unit: participants
Groups:
- No Intervention: Standard of Care: Patients will receive standard of care measures in case of cardiac arrest. They will not receive AECD monitoring or intervention.
Arm/Group | Experimental: AECD Monitoring + Standard of Care Group | No Intervention: Standard of Care
Number analyzed (Participants) | 95 | 97
participants | 95 | 97

4. Secondary Outcome: Cerebral Performance at Discharge
Description: Cerebral Performance Categories/CPC scale:
  CPC 1: Good cerebral performance - conscious, alert, able to work, might have mild neurologic or psychological deficit.
  CPC 2: Moderate cerebral disability - conscious, sufficient cerebral function for independent activities of daily life. Able to work in sheltered environment.
  CPC 3: Severe cerebral disability - conscious, dependent on others for daily support because of impaired brain function. Ranges from ambulatory state to severe dementia or paralysis.
  CPC 4: Coma or vegetative state - any degree of coma without the presence of all brain death criteria. Unawareness, even if appears awake (vegetative state) without interaction with environment; may have spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness.
  CPC 5: Brain death - apnea, areflexia, electroencephalogram (EEG) silence, etc.
Time Frame: At discharge
Population: Only 1 patient in the Intervention group had defibrillation during hospital admission and his CPC was 1.
Measure: Number; unit: units on a scale: CPC 1
Arm/Group | AECD Monitoring + Standard of Care Group | Standard of Care Group
Number analyzed (Participants) | 1 | 0
units on a scale: CPC 1 | 1 |

ADVERSE EVENTS:
Arm/Group | Experimental: AECD Monitoring + Standard of Care Group | No Intervention: Standard of Care Group
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/97
Other Adverse Events (participants affected / at risk) | 10/95 | 0/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: AECD Monitoring + Standard of Care Group (N=95) | No Intervention: Standard of Care Group (N=97)
False Positive Events in which, the shocks were delivered inappropriately. (Cardiac disorders) | 2 (2) | 0 (0) — 1. AECD delivered the shock when patient was eating an apple. 2. Discharge was the result of deliberate action of the patient.
Anxiety (Cardiac disorders) | 2 (2) | 0 (0)
Skin irritation by the pads (Cardiac disorders) | 2 (2) | 0 (0)
Alarming of the AECD, as the pads detached from the chest wall during sleep (Cardiac disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No